CLINICAL TRIAL: NCT05299359
Title: A Phase 3, Single Arm, Open-Label Trial to Evaluate the Immunogenicity and Safety of a Single Heterologous Booster Vaccination of TAK-019 in Healthy Japanese Male and Female Adults Aged 20 Years and Older (COVID-19)
Brief Title: A Single Heterologous Booster Vaccination Study of TAK-019 in Healthy Japanese Adults (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TAK-019-3001; jRCT2071210141 (Registry Identifier: jRCT); U1111-1281-3948 (Other: WHO)
Record Dates: First submitted 2022-03-27; First posted 2022-03-29 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAK-019 Main Part (Experimental): TAK-019 0.5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm
  Interventions: Biological: TAK-019
- TAK-019 Extension Part (Experimental): TAK-019 0 .5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm. The participants who received the first single booster vaccination of TAK-019 in the main part and remained in study follow-up at least 5 months will receive a second single booster vaccination of TAK-019 by intramuscular injection.
  Interventions: Biological: TAK-019

INTERVENTIONS:
Biological: TAK-019 — TAK-019 intramuscular injection

SUMMARY:
TAK-019 is a vaccine in development to protect people against Covid-19. The main aims of the study are to learn if TAK-019 can protect people from Covid-19 and to check for side effects from TAK-019 for participants who will receive TAK-019 as heterologous booster vaccination.

This study consists of two parts, main part and extension part. Firstly, participants who completed 2 doses primary vaccinations 6 to 12 months prior to the trial vaccination can take part in main study. At the first visit of main part of this study, the study doctor will check if each person can take part. Participants who can take part will receive an injection of TAK-019 as booster vaccination.

Participants will be asked to record their temperature and any medical problems in an electronic diary for up to 7 days after the injection. During the main part, participants will visit the clinic for regular check-ups, blood tests, and sometimes for nose swab samples. When all participants have attended a clinic visit 28 days after the injection, the study sponsor (Takeda) will check how many participants have made enough antibodies to protect them against Covid-19.

Participants who received the first single booster vaccination of TAK-019 in the main part and remained in study follow-up at least 5 months will be able to decide to take part in the extension part of this study. At the first visit of extension part of this study, the study doctor will check if each person can take part. Participants who can take part will receive an injection of TAK-019 as a second booster vaccination at the first visit of extension part.

The participants will stay in the main part of this study for up to 12 months after they have had their injection or up to the start of extension part. For participants who will take part in the extension part, they will stay in the extension part for up to 12 months from the start of extension part. During this time, the doctors will continue to collect blood samples to check immune response. Also, they will check if participants have any more side effects from TAK-019.

ELIGIBILITY:
Inclusion Criteria:

MAIN PART:

1. Healthy Japanese male and female adult participants aged >= 20 years of age at the time of signing of informed consent.
2. Participant who completed 2 doses primary vaccinations with another specified mRNA vaccine which is available in Japan 6 to 12 months prior to the trial vaccination.

   EXTENSION PART:
3. Participants who received the first trial vaccination at least 5 months earlier and are currently enrolled in the Main Part (ie, not have withdrawn or discontinued early).

Exclusion Criteria:

MAIN PART:

1. Participants who received any other SARS-CoV-2 vaccine (except for the specified mRNA vaccine) or other experimental novel coronavirus vaccine prior to the trial.
2. Participant who received a booster vaccination (i.e. 3rd dose)
3. Participants who have close contact of anyone known to have COVID-19 within 14 days prior to the trial vaccination.
4. Participants who were tested positive for SARS-CoV-2 prior to the trial.
5. Participants who have traveled outside of Japan in the 30 days prior to the trial participation.
6. Participants with a clinically significant active infection or oral temperature >= 38 degree Celsius within 3 days of the intended date of the first single booster vaccination.
7. Participants with body mass index (BMI) greater than or equal to 30 kg/m^2 (BMI= weight in kg/ height in meters^2)

   EXTENSION PART:
8. Participants with a clinically significant active infection or oral temperature >=38 degree Celsius within 3 days of the intended date of the second single booster vaccination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Sumida Hospital, Sumida-ku, Tokyo
  - PS Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kuriyama K, Murakami K, Sugiura K, Sakui S, Schuring RP, Mori M. Immunogenicity and safety of a second heterologous booster dose of NVX-CoV2373 (TAK-019) in healthy Japanese adults who had previously received a primary series of COVID-19 mRNA vaccine: Interim analysis report of a phase 3 open-label trial. Vaccine. 2024 Jan 25;42(3):662-670. doi: 10.1016/j.vaccine.2023.12.036. Epub 2023 Dec 21. PMID 38129286
- [Derived] Kuriyama K, Murakami K, Masuda T, Sugiura K, Sakui S, Schuring RP, Mori M. Immunogenicity and safety of a single booster dose of NVX-CoV2373 (TAK-019) in healthy Japanese adults who had previously received a primary series of COVID-19 mRNA vaccine: Primary analysis report of a phase 3 open-label trial. Vaccine. 2023 Jun 7;41(25):3763-3771. doi: 10.1016/j.vaccine.2023.05.001. Epub 2023 May 8. PMID 37198021
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/234514379776426d?id=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan. Healthy Japanese participants who completed 2 doses of primary vaccinations 6 to 12 months prior to trial vaccination were enrolled to receive a first dose of single booster vaccination of TAK-019 in Main Part and a second dose of booster vaccination of TAK-019 in Extension Part.
Pre-assignment Details: Participants were followed for up to 12 months after each vaccination in both parts. However, participants who remained for at least 5 months in Main Part were offered second single booster vaccination of TAK-019 in Extension Part, leading to a total participation duration of approximately 17 months.
Groups:
- Main Part: TAK-019: Participants received a first single booster vaccination of TAK-019 0.5 milliliter (mL), intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm at Day 1 of Main Part.
- Extension Part: TAK-019: Participants received a second booster vaccination of TAK-019 0.5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm at Day 1 of Extension Part.
Period: Main Part: Day 1 up to Day 366
Arm/Group | Main Part: TAK-019 | Extension Part: TAK-019
Started | 150 | 0
Completed | 17 | 0
Not Completed | 133 | 0
Not completed — Participants moved to extension part | 129 | 0
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Extension Part: Day 1 to Day 366
Arm/Group | Main Part: TAK-019 | Extension Part: TAK-019
Started | 0 | 129 (Participants who had received the first single booster vaccination of TAK-019 in the Main Part and remained in study follow-up for at least 5 months were offered second single booster vaccination of TAK-019 in Extension Part.)
Completed | 0 | 121
Not Completed | 0 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of the trial vaccination.
Groups:
- Main Part: TAK-019: Participants received a first single booster vaccination of TAK-019 0.5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm at Day 1 of Main Part.
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 150
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 150
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 61.70 (11.497)
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 164.47 (9.408)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] | 22.68 (2.940)

OUTCOME MEASURES:

1. Primary Outcome: Main Part: Geometric Mean Titers (GMT) Ratio of Neutralizing Antibody Titers to the Ancestral Strain (Wild-type Virus) on Day 15 Compared With That Observed on Day 36 in Participants From the TAK-019-1501 Study
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values was measured as below lower limit of quantification (LLOQ) were imputed to a value that was half of the LLOQ. LLOQ was equal to 20. GMT for each group and GMT ratio of neutralizing antibody titers to the ancestral strain (wild-type virus) on Day15 after a single booster vaccination (14 days after the booster vaccination) compared with that observed on Day 36 (14 days after the second vaccination) in participants from the TAK-019-1501 study (NCT04712110) were reported. GMT ratio was calculated with GMT of TAK-019-3001 on Day 15 divided by GMT of TAK-019-1501 study on Day 36. Here, ELISA is Enzyme-linked immunosorbent assay.
Time Frame: Day 15 for this study (14 days after the vaccination); Day 36 for TAK-019-1501 study (14 days after the second vaccination)
Population: Per-protocol Set: PPS was defined to include participants in the Full Analysis Set (FAS) and who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment. FAS was defined as all enrolled participants who received at least 1 dose of the trial vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per mL (EU/mL)
Groups:
- Main Part: Day 15 of This Study: TAK-019: Participants received a first single booster vaccination of TAK-019 0.5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm at Day 1 of Main Part.
- Day 36 for TAK-019-1501 Study: TAK-019 0.5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm, once on Days 1 and 22.
Arm/Group | Main Part: Day 15 of This Study: TAK-019 | Day 36 for TAK-019-1501 Study
Number analyzed (Participants) | 148 | 150
ELISA units per mL (EU/mL) | 1143.9 [1000.5 to 1307.9] | 884.4 [749.0 to 1044.4]
Statistical Analysis 1: Comparison: Main Part: Day 15 of This Study: TAK-019 vs Day 36 for TAK-019-1501 Study; GMT ratio was calculated GMT of TAK-019-3001 on Day 15 divided by GMT of TAK-019-1501 study on Day 36; Test type: Non-Inferiority — If the lower limit of the 95% CI is >= 0.67, then the immune response to a single heterologous booster vaccination of TAK-019 is considered to be non-inferior of that to the primary series of TAK-019; LS Mean Difference = 1.18, 95% CI 2-sided [0.95 to 1.47]

2. Primary Outcome: Main Part: Percentage of Participants With Reported Solicited Local Adverse Events (AEs) for 7 Days Following the First Single Booster Vaccination
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant administered an investigational medicinal product (IMP); it did not necessarily have to have a causal relationship with IMP administration. Reported solicited local AEs were defined as injection site pain, tenderness, erythema/redness, induration, and swelling.
Time Frame: Main Part: 7 days after the first single booster vaccination
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of the trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 74.0

3. Primary Outcome: Main Part: Percentage of Participants With Solicited Systemic AEs for 7 Days Following the First Single Booster Vaccination
Description: Solicited systemic AEs were defined as fever, fatigue, malaise, myalgia, arthralgia, nausea/vomiting, and headache.
Time Frame: Main Part: 7 days after the first single booster vaccination
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of the trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 48.0

4. Primary Outcome: Main Part: Percentage of Participants With Unsolicited AEs for 28 Days Following the First Single Booster Vaccination
Description: Unsolicited AEs defines as other AEs than solicited local AEs and solicited systemic AEs.
Time Frame: Main Part: 28 days after the first single booster vaccination
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 4.67

5. Primary Outcome: Main Part: Percentage of Participants With Solicited and Unsolicited Serious Adverse Events (SAE) Until Day 29
Description: An SAE was defined as any untoward medical occurrence that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or is an important medical event. Solicited SAEs and unsolicited SAEs were reported.
Time Frame: Main Part: Up to Day 29
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants
  Solicited SAEs up to Day 29 | 0
  Unsolicited SAEs up to Day 29 | 0

6. Primary Outcome: Main Part: Percentage of Participants With Adverse Event of Special Interest (AESI) Until Day 29
Description: An AESI was defined as AEs that will be specifically highlighted to the Investigator. AESIs for the study included the Potential Immune Mediated Medical Conditions (PIMMC) and AEs specific to COVID-19. PIMMC is categorized as following; neuroinflammatory disorders, musculoskeletal and connective tissue disorders, vasculitides, gastrointestinal disorders, hepatic disorders, renal disorders, cardiac disorders, skin disorder, hematologic disorders, metabolic disorders, and other disorders.
Time Frame: Main Part: Up to Day 29
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 0

7. Primary Outcome: Main Part: Percentage of Participants With Medically-Attended Adverse Events (MAAEs) Until Day 29
Description: MAAEs were defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: Main Part: Up to Day 29
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 0.7

8. Primary Outcome: Main Part: Percentage of Participants With Any AE Leading to Withdrawal From the Trial Until Day 29
Description: Percentage of participants with any AE leading to withdrawal from the trial until Day 29 was reported.
Time Frame: Main Part: Up to Day 29
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 0

9. Primary Outcome: Main Part: Percentage of Participants With Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Infection Until Day 29
Description: Percentage of participants with SARS-CoV-2 infection until Day 29 of the main part of the trial were reported in this outcome measure.
Time Frame: Main Part: Up to Day 29
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
Percentage of Participants | 0

10. Secondary Outcome: Main Part: GMT of Serum Immunoglobulin G (IgG) Antibody Levels to SARS-CoV-2 Recombinant Spike (rS) Protein on Day 8, 15, 29, 91, 181, and 366
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average. Titer values was measured as below LLOQ were imputed to a value that was half of the LLOQ. LLOQ was equal to 200 EU/mL.
Time Frame: Main Part: Day 8, 15, 29, 91, 181, and 366
Population: Per-protocol Set: PPS was defined to include participants in the FAS and who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment. Here, "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 148
EU/mL
  At Day 8 | 24705.9 [21894.6 to 27878.2]
  At Day 15 | 35202.2 [31508.4 to 39329.1]
  At Day 29 | 36138.3 [32143.8 to 40629.2]
  At Day 91: number analyzed (Participants) | 139
  At Day 91 | 26420.8 [23137.2 to 30170.4]
  At Day 181: number analyzed (Participants) | 15
  At Day 181 | 20246.3 [11976.5 to 34226.5]
  At Day 366: number analyzed (Participants) | 13
  At Day 366 | 31369.4 [15135.7 to 65014.5]

11. Secondary Outcome: Main Part: Geometric Mean Fold Rise (GMFR) of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Day 8, 15, 29, 91, 181, and 366
Description: GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Where baseline was defined as the last measurement taken before the first dose of trial vaccination.
Time Frame: Main Part: Day 8, 15, 29, 91, 181, and 366
Population: Per-protocol Set: PPS was defined to include participants in the FAS and who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment. Here, number analyzed signifies participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 148
fold rise
  At Day 8 | 4.21 [3.69 to 4.81]
  At Day 15 | 6.00 [5.17 to 6.97]
  At Day 29 | 6.16 [5.23 to 7.27]
  At Day 91: number analyzed (Participants) | 139
  At Day 91 | 4.43 [3.67 to 5.36]
  At Day 181: number analyzed (Participants) | 15
  At Day 181 | 2.96 [1.45 to 6.04]
  At Day 366: number analyzed (Participants) | 13
  At Day 366 | 4.28 [1.33 to 13.77]

12. Secondary Outcome: Main Part: Seroconversion Rate (SCR) of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Day 8, 15, 29, 91, 181, and 366
Description: SCR was defined as percentage of participants with 4-fold or more rises from baseline in titer. Baseline was defined as the last measurement taken before the first dose of trial vaccination.
Time Frame: Main Part: Day 8, 15, 29, 91, 181, and 366
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 148
percentage of participants
  At Day 8 | 53.4 [45.0 to 61.6]
  At Day 15 | 70.9 [62.9 to 78.1]
  At Day 29 | 70.3 [62.2 to 77.5]
  At Day 91: number analyzed (Participants) | 139
  At Day 91 | 56.1 [47.5 to 64.5]
  At Day 181: number analyzed (Participants) | 15
  At Day 181 | 40.0 [16.3 to 67.7]
  At Day 366: number analyzed (Participants) | 13
  At Day 366 | 61.5 [31.6 to 86.1]

13. Secondary Outcome: Main Part: GMT of Serum Neutralizing Antibody Titers to the Ancestral Strain (Wild-type Virus) on Day 8, 15, 29, 91, 181, and 366
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which greater than or equal to (>=) 50 percent (%) of the replicate wells were protected from infection (microneutralization [MN] with an inhibitory concentration of 50% [MN50]). GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average. Titer values was measured as below LLOQ were imputed to a value that was half of the LLOQ where LLOQ was equal to 20.
Time Frame: Main Part: Day 8, 15, 29, 91, 181, and 366
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: 1 per dilution
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 148
1 per dilution
  At Day 8 | 729.7 [634.5 to 839.2]
  At Day 15 | 1143.9 [1000.5 to 1307.9]
  At Day 29 | 775.5 [693.8 to 866.8]
  At Day 91: number analyzed (Participants) | 139
  At Day 91 | 656.2 [559.6 to 769.4]
  At Day 181: number analyzed (Participants) | 15
  At Day 181 | 844.5 [410.0 to 1739.3]
  At Day 366: number analyzed (Participants) | 13
  At Day 366 | 1424.0 [597.0 to 3396.9]

14. Secondary Outcome: Main Part: GMFR of Serum Neutralizing Antibody Titers to the Ancestral Strain (Wild-type Virus) on Day 8, 15, 29, 91, 181, and 366
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which >=50% of the replicate wells were protected from infection (MN50). GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Baseline was defined as the last measurement taken before the first dose of trial vaccination.
Time Frame: Main Part: Day 8, 15, 29, 91, 181, and 366
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 148
fold rise
  At Day 8 | 5.32 [4.55 to 6.23]
  At Day 15 | 8.34 [6.93 to 10.04]
  At Day 29 | 5.66 [4.68 to 6.84]
  At Day 91: number analyzed (Participants) | 139
  At Day 91 | 4.72 [3.72 to 5.97]
  At Day 181: number analyzed (Participants) | 15
  At Day 181 | 5.79 [2.43 to 13.80]
  At Day 366: number analyzed (Participants) | 13
  At Day 366 | 9.90 [2.84 to 34.54]

15. Secondary Outcome: Main Part: SCR of Serum Neutralizing Antibody Titters to the Ancestral Strain (Wild-type Virus) on Day 8, 15, 29, 91, 181, and 366
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which greater than or equal to (>=) 50% of the replicate wells were protected from infection (MN50). SCR was defined as percentage of participants with 4-fold or more rises in from baseline. Baseline was defined as the last measurement taken before the first dose of trial vaccination.
Time Frame: Main Part: Day 8, 15, 29, 91, 181, and 366
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 148
percentage of participants
  At Day 8 | 77.7 [70.1 to 84.1]
  At Day 15 | 84.5 [77.6 to 89.9]
  At Day 29 | 75.7 [67.9 to 82.3]
  At Day 91: number analyzed (Participants) | 139
  At Day 91 | 67.6 [59.2 to 75.3]
  At Day 181: number analyzed (Participants) | 15
  At Day 181 | 66.7 [38.4 to 88.2]
  At Day 366: number analyzed (Participants) | 13
  At Day 366 | 76.9 [46.2 to 95.0]

16. Secondary Outcome: Main Part: Percentage of Participants With Solicited and Unsolicited SAEs Throughout the Main Part of Trial
Description: as for outcome 5
Time Frame: Main Part: Up to Day 366
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
percentage of participants
  Solicited SAEs Throughout the Main Part of Trial | 0
  Unsolicited SAEs Throughout the Main Part of Trial | 0

17. Secondary Outcome: Main Part: Percentage of Participants With AESI Throughout the Main Part of Trial
Description: An AESI was defined as AEs that will be specifically highlighted to the Investigator. AESIs for the study included the PIMMC and AEs specific to COVID-19. PIMMC is categorized as following; neuroinflammatory disorders, musculoskeletal and connective tissue disorders, vasculitides, gastrointestinal disorders, hepatic disorders, renal disorders, cardiac disorders, skin disorder, hematologic disorders, metabolic disorders, and other disorders.
Time Frame: Main Part: Up to Day 366
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
percentage of participants | 0

18. Secondary Outcome: Main Part: Percentage of Participants With MAAEs Throughout the Main Part of Trial
Description: as for outcome 7
Time Frame: Main Part: Up to Day 366
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
percentage of participants | 20.0

19. Secondary Outcome: Main Part: Percentage of Participants With Any AE Leading to Participant's Withdrawal From the Trial From the Day of the First Single Booster Vaccination Throughout the Main Part of Trial
Description: Percentage of participants with any AE leading to participant's withdrawal from the trial from the day of the first single booster vaccination throughout the main part of trial was reported.
Time Frame: Main Part: Day 1 up to Day 366
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of the trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
percentage of participants | 0

20. Secondary Outcome: Main Part: Percentage of Participants With SARS-CoV-2 Infection Throughout the Main Part of Trial
Description: Percentage of participants with SARS-CoV-2 infection throughout the main part of trial was reported.
Time Frame: Main Part: Day 1 up to Day 366
Population: Main Part: The safety analysis set included all participants who received at least 1 dose of the trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Main Part: TAK-019
Number analyzed (Participants) | 150
percentage of participants | 14.0

21. Secondary Outcome: Extension Part: GMT of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Day 15, 29, 91, 181, and 366
Description: as for outcome 10
Time Frame: Extension Part: Day 15, 29, 91, 181, and 366
Population: Extension Part PPS was defined to include participants in the FAS in the Extension Part who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment. Here, "overall number of participants analyzed" signified participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Groups:
- Extension Part: TAK-019: Participants received TAK-019 0.5 mL, intramuscular injection in the mid deltoid, preferable in the non-dominant upper arm at Day 1 of Extension part.
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 111
EU/mL
  At Day 15 | 105057.6 [91624.1 to 120460.6]
  At Day 29: number analyzed (Participants) | 110
  At Day 29 | 88154.1 [77487.0 to 100289.7]
  At Day 91: number analyzed (Participants) | 107
  At Day 91 | 61090.0 [52488.3 to 71101.2]
  At Day 181: number analyzed (Participants) | 102
  At Day 181 | 46199.1 [38752.6 to 55076.6]
  At Day 366: number analyzed (Participants) | 90
  At Day 366 | 62823.7 [51897.3 to 76050.6]

22. Secondary Outcome: Extension Part: GMFR of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Extension Part Day 15, 29, 91, 181, and 366
Description: The GMFR was calculated as the ratio of the post-second-booster-vaccination titer level to extension part baseline titer level. Where extension part baseline was defined as last measurement taken before the second booster vaccination.
Time Frame: Extension Part: Day 15, 29, 91, 181, and 366
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 111
fold rise
  At Day 15 | 3.99 [3.47 to 4.59]
  At Day 29: number analyzed (Participants) | 110
  At Day 29 | 3.32 [2.91 to 3.78]
  At Day 91: number analyzed (Participants) | 107
  At Day 91 | 2.30 [1.96 to 2.70]
  At Day 181: number analyzed (Participants) | 102
  At Day 181 | 1.72 [1.43 to 2.08]
  At Day 366: number analyzed (Participants) | 90
  At Day 366 | 2.33 [1.84 to 2.95]

23. Secondary Outcome: Extension Part: Seroconversion Rate (SCR) of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Extension Part Day 15, 29, 91, 181, and 366
Description: SCR was defined as percentage of participants with 4-fold or more rises in titer from extension part baseline. Where extension part baseline was defined as last measurement taken before the second booster vaccination.
Time Frame: Extension Part: Day 15, 29, 91, 181, and 366
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 111
percentage of participants
  At Day 15 | 51.4 [41.7 to 61.0]
  At Day 29: number analyzed (Participants) | 110
  At Day 29 | 40.9 [31.6 to 50.7]
  At Day 91: number analyzed (Participants) | 107
  At Day 91 | 19.6 [12.6 to 28.4]
  At Day 181: number analyzed (Participants) | 102
  At Day 181 | 16.7 [10.0 to 25.3]
  At Day 366: number analyzed (Participants) | 90
  At Day 366 | 28.9 [19.8 to 39.4]

24. Secondary Outcome: Extension Part: GMT of Serum Neutralizing Antibody Titers to the Ancestral Strain (Wild-type Virus) on Extension Part Day 15, 29, 91, 181, and 366
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at >= 50% of the replicate wells were protected from infection (MN50). GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average. Titer values was measured as below LLOQ were imputed to a value that was half of the LLOQ where LLOQ was equal to 20.
Time Frame: Extension Part: Day 15, 29, 91, 181, and 366
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: 1 per dilution
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 111
1 per dilution
  At Day 15 | 1716.6 [1463.2 to 2013.9]
  At Day 29: number analyzed (Participants) | 110
  At Day 29 | 1732.1 [1465.8 to 2046.8]
  At Day 91: number analyzed (Participants) | 107
  At Day 91 | 1255.4 [1019.2 to 1546.3]
  At Day 181: number analyzed (Participants) | 102
  At Day 181 | 1360.7 [1081.2 to 1712.6]
  At Day 366: number analyzed (Participants) | 90
  At Day 366 | 660.0 [531.0 to 820.4]

25. Secondary Outcome: Extension Part: GMFR of Serum Neutralizing Antibody Titers to the Ancestral Strain (Wild-type Virus) on Extension Part Day 15, 29, 91, 181, and 366
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at >= 50% of the replicate wells were protected from infection (MN50). The GMFR was calculated as the ratio of the post-second-booster-vaccination titer level to extension part baseline titer level. Where extension part baseline was defined as last measurement taken before the second booster vaccination.
Time Frame: Extension Part: Day 15, 29, 91, 181, and 366
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 111
fold rise
  At Day 15 | 3.04 [2.59 to 3.57]
  At Day 29: number analyzed (Participants) | 110
  At Day 29 | 3.05 [2.57 to 3.63]
  At Day 91: number analyzed (Participants) | 107
  At Day 91 | 2.19 [1.81 to 2.66]
  At Day 181: number analyzed (Participants) | 102
  At Day 181 | 2.34 [1.86 to 2.94]
  At Day 366: number analyzed (Participants) | 90
  At Day 366 | 1.16 [0.86 to 1.55]

26. Secondary Outcome: Extension Part: SCR of Serum Neutralizing Antibody Titers to the Ancestral Strain (Wild-type Virus) on Extension Part Day 15, 29, 91, 181, and 366
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at >= 50% of the replicate wells were protected from infection (MN50). SCR was defined as percentage of participants with 4-fold or more rises in titer from extension part baseline.
Time Frame: Extension Part: Day 15, 29, 91, 181, and 366
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 111
percentage of participants
  At Day 15 | 51.4 [41.7 to 61.0]
  At Day 29: number analyzed (Participants) | 110
  At Day 29 | 52.7 [43.0 to 62.3]
  At Day 91: number analyzed (Participants) | 107
  At Day 91 | 30.8 [22.3 to 40.5]
  At Day 181: number analyzed (Participants) | 102
  At Day 181 | 36.3 [27.0 to 46.4]
  At Day 366: number analyzed (Participants) | 90
  At Day 366 | 24.4 [16.0 to 34.6]

27. Secondary Outcome: Extension Part: Percentage of Participants With Reported Solicited Local AEs for 7 Days Following the Second Single Booster Vaccination in Extension Part
Description: as for outcome 2
Time Frame: Extension Part: 7 days after the second single booster vaccination
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 73.6

28. Secondary Outcome: Extension Part: Percentage of Participants With Solicited Systemic AEs for 7 Days Following the Second Single Booster Vaccination in Extension Part
Description: Solicited systemic AEs included were defined as fever, fatigue, malaise, myalgia, arthralgia, nausea/vomiting and headache.
Time Frame: Extension Part: 7 days after the second single booster vaccination
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 51.2

29. Secondary Outcome: Extension Part: Percentage of Participants With Unsolicited AEs for 28 Days Following the Second Single Booster Vaccination in Extension Part
Description: Unsolicited AEs defined as AEs other than solicited local AEs and solicited systemic AEs.
Time Frame: Extension Part: 28 days after the second single booster vaccination
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 7.0

30. Secondary Outcome: Extension Part: Percentage of Participants With Solicited and Unsolicited SAEs Until Extension Part Day 29
Description: as for outcome 5
Time Frame: Extension Part: Up to Day 29
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants
  Solicited SAEs Up to Extension Part Day 29 | 0
  Unsolicited SAEs Up to Extension Part Day 29 | 0.8

31. Secondary Outcome: Extension Part: Percentage of Participants With AESIs Until Extension Part Day 29
Description: as for outcome 17
Time Frame: Extension Part: Up to Day 29
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 0

32. Secondary Outcome: Extension Part: Percentage of Participants With MAAEs Until Extension Part Day 29
Description: as for outcome 7
Time Frame: Extension Part: Up to Day 29
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 5.4

33. Secondary Outcome: Extension Part: Percentage of Participants With Any AEs Leading to Withdrawal From the Trial Until Extension Part Day 29
Description: Percentage of participants with any AEs leading to withdrawal from the trial until extension part Day 29 was reported.
Time Frame: Extension Part: Up to Day 29
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 0

34. Secondary Outcome: Extension Part: Percentage of Participants With SARS-CoV-2 Infection Until Extension Part Day 29
Description: Percentage of participants with SARS-CoV-2 infection until extension part Day 29 was reported.
Time Frame: Extension Part: Up to Day 29
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 0

35. Secondary Outcome: Extension Part: Percentage of Participants With Solicited and Unsolicited SAEs Throughout the Extension Part of the Trial
Description: as for outcome 5
Time Frame: Extension Part: Up to Day 366
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants
  Solicited SAEs Throughout the Extension Part | 0
  Unsolicited SAEs Throughout the Extension Part | 3.1

36. Secondary Outcome: Extension Part: Percentage of Participants With AESIs Throughout the Extension Part of the Trial
Description: as for outcome 17
Time Frame: Extension Part: Up to Day 366
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 0

37. Secondary Outcome: Extension Part: Percentage of Participants With MAAEs Throughout the Extension Part of the Trial
Description: as for outcome 7
Time Frame: Extension Part: Up to Day 366
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 31.0

38. Secondary Outcome: Extension Part: Percentage of Participants With Any AEs Leading to Withdrawal From the Trial From the Day of the Second Single Booster Vaccination Throughout the Extension Part of the Trial
Description: Percentage of participants with any AEs leading to withdrawal from the trial from the day of the second single booster vaccination throughout the extension part of the trial was reported.
Time Frame: Extension Part: From Day 1 up to Day 366
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 0

39. Secondary Outcome: Extension Part: Percentage of Participants With SARS-CoV-2 Infection Throughout the Extension Part of Trial
Description: Percentage of participants with SARS-CoV-2 infection throughout the extension part of trial was reported.
Time Frame: Extension Part: Up to Day 366
Population: Extension Part: The safety analysis set included all participants who received at least 1 dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Part: TAK-019
Number analyzed (Participants) | 129
percentage of participants | 10.9

ADVERSE EVENTS:
Time Frame: Main Part: Day 1 up to 366 and Extension Part: Day 1 up to Day 366 (Participants who participated in the Main Part and the Extension Part, total participation duration was approximately 17 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Main Part: TAK-019 | Extension Part: TAK-019
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/150 | 4/129
Other Adverse Events (participants affected / at risk) | 123/150 | 107/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Part: TAK-019 (N=150) | Extension Part: TAK-019 (N=129)
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Part: TAK-019 (N=150) | Extension Part: TAK-019 (N=129)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 18
COVID-19 (Infections and infestations) | 21 | 14
Fatigue (General disorders) | 28 | 33
Headache (Nervous system disorders) | 37 | 37
Injection site pain (General disorders) | 80 | 65
Malaise (General disorders) | 39 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 29 | 34
Nasopharyngitis (Infections and infestations) | 1 | 10
Nausea (Gastrointestinal disorders) | 10 | 11
Swelling (General disorders) | 7 | 11
Tenderness (General disorders) | 102 | 89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT05299359/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05299359/SAP_002.pdf